CLINICAL TRIAL: NCT05180929
Title: The Comparative Effects of Dual-tDCS and Anodal Premotor tDCS Over the Contralesional Hemisphere on the Upper Limb Function and Manual Dexterity in Patients With Chronic Stroke: Single-blinded Randomized Controlled Trial
Brief Title: Dual-tDCS and Anodal PMC tDCS Over the Contralesional Hemisphere on the Upper Limb Function in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turki Abualait (Other Government)
Responsible Party: Sponsor-Investigator, Turki Abualait, Chair of Physical Therapy Department, Assistant Professor of Cognitive Neuroscience and Neurorehabilitation, Imam Abdulrahman Al Faisal Hospital
Organization: Imam Abdulrahman Al Faisal Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IAU
Record Dates: First submitted 2021-11-16; First posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Stroke
Keywords: tDCS; PMC; IHI; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Dual-M1 tDCS (Experimental): In the M1- dual tDCS montage, the anodal electrode will be placed above ipsilesional M1 and the cathode will be positioned over contralesional M1.
  Interventions: Device: Dual M1-tDCS
- a-tDCS over contralesional PMC (Experimental): In the anodal-tDCS for PMC, the anodal electrode will be placed over the contralesional PMC. The PMC is defined as being 2.5 cm anterior to the M1. The cathodal electrode will be positioned over the contralateral suborbital region
  Interventions: Device: a-tDCS over contralesional PMC
- Sham tDCS (Sham Comparator): For sham stimulation, there is no particular electrode configuration to be followed, thus, 6 participants will receive sham stimulation with the configuration will be used in group A, and 5 participants will receive sham stimulation with the configuration will be used in group B. By pressing the sham button, the current will automatically ramped up over 10 sec. till reaching 1 mA, then it will be decreased gradually over 30 seconds till turning off the apparatus. This is to ensure the typical initial itching sensation
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Dual M1-tDCS — In the M1- dual tDCS montage, the anodal electrode will be placed above ipsilesional M1 and the cathode will be positioned over contralesional M1.
  Arms: Dual-M1 tDCS
Device: a-tDCS over contralesional PMC — In the anodal-tDCS for PMC, the anodal electrode will be placed over the contralesional PMC. The PMC is defined as being 2.5 cm anterior to the M1. The cathodal electrode will be positioned over the contralateral suborbital region
  Arms: a-tDCS over contralesional PMC
Device: Sham tDCS — For sham stimulation, there is no particular electrode configuration to be followed, thus, 6 participants will receive sham stimulation with the configuration will be used in group A, and 5 participants will receive sham stimulation with the configuration will be used in group B. By pressing the sham button, the current will automatically ramped up over 10 sec. till reaching 1 mA, then it will be decreased gradually over 30 seconds till turning off the apparatus. This is to ensure the typical initial itching sensation
  Arms: Sham tDCS

SUMMARY:
Background: Transcranial direct current stimulation (tDCS) has been gaining increasing interest as a potential therapeutic tool to improve upper extremity (UE) rehabilitation outcomes following stroke. Within the concept of interhemispheric inhibition (IHI), most tDCS studies have applied anodal ipsilesional and/or cathodal contralesional primary motor cortex (M1) tDCS to rebalance IHI and enhance motor recovery. However, compelling evidence suggests that an excitation/inhibition model is oversimplified, and the role of both hemispheres in the encoding of information during motor learning should be acknowledged. Moreover, multiple lines of evidence have demonstrated the potential relevance of contralesional premotor cortex (PMC) for recovery after M1 injury.

Objective: We are aiming to investigate and compare the eﬀects of two tDCS montages at different cortical sites (Dual-M1 vs. a-tDCS over contralesional PMC) by measuring the clinical outcomes of the most affected UE in patients with chronic subcortical stroke.

Methods: 35 participants will be randomly assigned to 1 of 3 groups (Group A received dual- M1 tDCS, Group B received a-tDCS over contralesional PMC, and Group C received sham stimulation). tDCS will be applied using intensity of 2 mA for 20 min. (5 times/week) for 2 consecutive weeks. Fugl-Meyer Assessment of the Upper Extremity (FMA-UE) and Action Research Arm Test (ARAT) will be used to quantify the UE functional motor ability. Box and Block Test (BBT) will be used for gross manual dexterity and Nine Hole Peg Test (NHPT) will be used to measure fine hand dexterity. All measurements will be taken pre-treatment (T0) and post-treatment (T1) immediately after the 10th session, then 4 weeks after the end of stimulation period (T2) to assess the long-term effects.

Expected results: This study would verify whether enhancing the motor cortical hyperexcitability in the contralesional hemisphere has a beneficial on recovery of the paretic hand, or regaining the balance of transcallosal inhibitory circuits between the motor areas in both hemispheres has more positive effects on the motor outcomes . This study would also provide a predictive approach to enable realistic rehabilitation goal-setting by identifying the proper tDCS montage for patients with stroke depending on their impairment level.

DETAILED DESCRIPTION:
This experimental study will be conducted in a sham-controlled, single-blinded randomized controlled design. The subjects will be recruited - by convenience sampling - from the outpatient population of different governmental hospitals in Eastern Province of Saudi Arabia. Neurologists, Physiatrists and Physical therapists will be contacted to recruit potential subjects and IRB-approved letter will be sent to them. The subjects will be screened to determine whether a potential participant is eligible to be enrolled in the study or not. Only the principal investigator (PI) will conduct the screening procedures, which include reviewing medical record, in-person interview and administration of Mini-Mental State Examination. All screening activities will take 15-20 min., and they will be performed in a private screening room. Enrollment will occur after verifying the eligibility and obtaining the signed written consent form. Participants will be enrolled in the study only if they met all the inclusion criteria, which are:

1. Male or Female participants aged ≥ 18
2. First ever, unilateral, ischemic, subcortical stroke in the territories supplied by the Middle Cerebral Artery (MCA) verified by brain imaging, at chronic stage (≥ 6 months).
3. Upper Extremity impairment verified by Fugl-Meyer Assessment-Upper Extremity (FMA-UE).
4. Mini Mental State Examination Score ≥ 24.

All the participants were receiving conventional physical therapy and occupational therapy sessions (1-2 times/week).

The Exclusion Criteria included the following:

1. History of epileptic seizures.
2. Pre-stroke motor impairment(s) affecting UE.
3. Presence of UE contractures or deformities.
4. Botulinum toxin to UE muscles in the last 6 months.
5. Presence of damaged skin on the scalp that would interfere with tDCS stimulation.
6. Individuals with metallic implant in the brain or medical devices (i.e., cardiac pacemaker, deep brain stimulator, cochlear implants).
7. Use of CNS-affecting drugs.
8. Additional neurological or psychiatric problem.
9. Pregnancy.

After enrollment, all participants will be scheduled to receive 10 sessions over two consecutive weeks (5 sessions/week). Each participant will be seen initially (1st visit) for about 90 min. to conduct all baseline measurements (T0), which will include clinical examinations using different standardized tests for upper limb function, and to conduct the experiment. The follow up sessions (8 sessions) will last for around 30 min. (10 min. for preparation and employing the electrodes + 20 min. for the stimulation). The 10th session will last for about 90 min. to carry out the measurement tests (T1) and to conduct the last stimulation session. The final visit will be scheduled to be 4 weeks after the 10th session to evaluate the long-term effects using the same measurement tests (T2).

All the participants will be blinded to the type of stimulation they received. The PI will take all the baseline measurements (T0), post-stimulation measurements immediately after the 10th session (T1), and long-term effects 4 weeks after the end of the stimulation period (T2). The PI will carry out all tDCS sessions as well.

All the participants will be randomly assigned, using opaque envelopes, to one of three groups:

* Group A (n=11) receive dual-tDCS
* Group B (n=13) receive a-tDCS over PMC in the contralesional hemisphere, and
* Group C (n=11) receive sham stimulation.

This study protocol has been approved by the IRB from the research ethics committee in Imam Abdulrahman Bin Faisal University.

ELIGIBILITY:
Inclusion Criteria:

1. First ever, unilateral, ischemic, subcortical stroke in the territories supplied by the Middle Cerebral Artery (MCA) verified by brain imaging, at chronic stage (≥ 6 months).
2. Upper Extremity impairment verified by Fugl-Meyer Assessment-Upper Extremity (FMA-UE)
3. Mini Mental State Examination Score ≥ 24

Exclusion Criteria:

1. History of epileptic seizures.
2. Pre-stroke motor impairment(s) affecting UE.
3. Presence of UE contractures or deformities.
4. Botulinum toxin to UE muscles in the last 6 months.
5. Presence of damaged skin on the scalp that would interfere with tDCS stimulation.
6. Individuals with metallic implant in the brain or medical devices (i.e., cardiac pacemaker, deep brain stimulator, cochlear implants).
7. Use of CNS-affecting drugs.
8. Additional neurological or psychiatric problem.
9. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-14 (Actual)

PRIMARY OUTCOMES:
Change from Baseline 'Fugl-Meyer Assessment of the Upper Extremity (FMA-UE)' at 4 weeks | T0: Baseline measurements (immediately prior stimulation), T1: Post-stimulation measurements (2 weeks after T0), T2: 4 weeks after T1 to evaluate the long-term effects
  the most frequently used outcome measure when assessing UE function after stroke within the research context (Santisteban et al., 2016). We will exclude the 3 reflex items because they make no difference to the overall scores of the test (Gladstone, Danells and Black, 2002; Woodbury et al., 2007; Woytowicz et al., 2017). It is composed of 30 items, each scored on a scale of 0 to 2. It has an excellent overall reliability (Duncan, Propst and Nelson, 1983; Sanford et al., 1993), validity and responsiveness as an indicator of motor impairment severity across different stroke recovery time points (Platz et al., 2005; Hsieh et al., 2009).

SECONDARY OUTCOMES:
Change from Baseline 'Action Research Arm Test (ARAT)' at 4 weeks | T0: Baseline measurements (immediately prior stimulation), T1: Post-stimulation measurements (2 weeks after T0), T2: 4 weeks after T1 to evaluate the long-term effects
  is a standardized, observational measure of UE functional capability for adult stroke survivors. It includes 19 items categorized into four subscales (grasp, grip, pinch and gross movement). Task performance on each item is rated on a 4-point ordinal scale, ranging from 0 (no movement) to 3 (movement performed normally) (Yozbatiran, Der-Yeghiaian and Cramer, 2008).
Change from Baseline 'Box and Block Test (BBT)' at 4 weeks | T0: Baseline measurements (immediately prior stimulation), T1: Post-stimulation measurements (2 weeks after T0), T2: 4 weeks after T1 to evaluate the long-term effects
  to assess gross manual dexterity. It consists of a wooden box divided by a partition into two equal compartments with 150 wooden blocks placed in one compartment. The participants will be given 60 seconds to move, one by one, as many 2.5 cm blocks as possible from one compartment to the other using only the most affected hand. 15-second trial will be allowed for each participant at the beginning to ensure adequate understanding of the task. BBT has excellent test-retest reliability when tested on more affected (r = 0.98) and less affected hand (r = 0.93) (Chen et al., 2009).
Change from Baseline 'Nine Hole Peg Test (NHPT)' at 4 weeks | T0: Baseline measurements (immediately prior stimulation), T1: Post-stimulation measurements (2 weeks after T0), T2: 4 weeks after T1 to evaluate the long-term effects
  is a finger dexterity measure involving timed performance to insert and remove 9 pegs from holes in a wooden board. It showed excellent test retest reliability (Chen et al., 2009), adequate to excellent intra-rater reliability and excellent inter-rater reliability (Heller et al., 1987).

CONTACTS AND LOCATIONS:
Locations (1):
- BrainStim Lab, Imam Abdulrahman Bin Faisal University, Dammam, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No